CLINICAL TRIAL: NCT05635370
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- Pentoxifylline Versus Cilostazol
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019P003607-12
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Pentoxifylline; Cilostazol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pentoxifylline: Exposure group
  Interventions: Drug: Pentoxifylline
- Cilostazol: Reference group
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline claim is used as the exposure group.
  Groups: Pentoxifylline
Drug: Cilostazol — Cilostazol claim is used as the reference group.
  Groups: Cilostazol

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/17QJ294pffmOCFYLeq0eSvn7hlj6MOb-0dJCr1RL3kfk/edit?usp=sharing or Appendix A (https://drive.google.com/drive/folders/1-lR6dR_aP44GoryjCad_NwRhjPpsIKDU?usp=sharing) for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability)

Inclusion Criteria:

* 1. Aged >/= 65 years on the index date
* 2. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 3. At least two claims with peripheral artery disease diagnosis measured 365 days prior to drug initiation

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior history of nursing home admission in the 365 days prior to the cohort entry date
* 3. Prior history of Pentoxifylline or Cilostazol use anytime prior to cohort entry date

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing Pentoxifylline versus Cilostazol. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 10398 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pentoxifylline | Cilostazol
Started | 1701 | 8697
Completed | 1687 | 1687
Not Completed | 14 | 7010

BASELINE CHARACTERISTICS:
Population: Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Cilostazol | Total
Number analyzed (Participants) | 1687 | 1687 | 3374
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1687 | 1687 | 3374
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.2 (7.2) | 76.1 (7.3) | 76.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 869 | 848 | 1717
  Male | 818 | 839 | 1657
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1378 | 1390 | 2768
  Black | 156 | 151 | 307
  Hispanic | 67 | 66 | 133
  Other | 86 | 80 | 166
Dementia risk factors [Count of Participants; unit: Participants]
  Anxiety | 244 | 242 | 486
  Bipolar Disorder | 15 | 18 | 33
  Coronary Artery Disease | 793 | 767 | 1560
  Depression | 236 | 243 | 479
  Diabetes | 819 | 807 | 1626
  Hypertension | 1501 | 1521 | 3022
  Obesity | 320 | 298 | 618

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.
Time Frame: Median follow up times: 1) 180 days (exp), 170 days (ref) 2) 677 days (exp), 612 days (ref) 3) 211 days (exp), 173 days (ref) 4) 180 days (exp), 171 days (ref)
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | Pentoxifylline | Cilostazol
Number analyzed (Participants) | 1687 | 1687
Incidence rate per 1000 person year
  Analysis 1 | 28.1 [20.2 to 38.2] | 32.6 [23.5 to 44.0]
  Analysis 2 | 37.9 [28.4 to 49.6] | 44.8 [34.2 to 57.7]
  Analysis 3 | 30.8 [18.8 to 47.6] | 43.9 [28.9 to 63.9]
  Analysis 4 | 5.2 [2.3 to 10.3] | 10.0 [5.3 to 17.2]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 180 (for Pentoxifylline) and 170 (for Cilostazol)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | Pentoxifylline | Cilostazol
All-Cause Mortality (participants affected / at risk) | 0/1687 | 0/1687
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1687 | 0/1687

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT05635370/Prot_SAP_000.pdf